CLINICAL TRIAL: NCT02419937
Title: Short-Term Application of Tocilizumab Following Myocardial Infarction
Acronym: STAT-MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FKE20140029H
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocilizumab (Active Comparator): Blinded subjects will be randomized to tocilizumab 162 mg subcutaneously once.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): Blinded subjects will be randomized to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — 162 mg subcutaneously once (vs. 0.9% normal saline placebo injection once in placebo arm)
  Other Names: Actemra
  Arms: Tocilizumab
Drug: Placebo — Saline injection
  Arms: Placebo

SUMMARY:
Introduction: Interleukin 6 (IL-6) is a cytokine that has a pro-inflammatory effect on the immune system. In acute MI IL-6 levels rapidly increase in response to ischemia and inflammation. Tocilizumab is a humanized monoclonal antibody against the interleukin-6 receptor (IL-6R). The use of tocilizumab within the first 24 hours of admission for acute MI could reduce 30 day mortality.

Methods: This randomized, placebo controlled trial will assign subjects within 24 hours of admission to treatment with either 162 mg of tocilizumab subcutaneously once or placebo in addition to usual pharmacologic and interventional standard of care for acute MI (ST segment elevation MI or non-ST segment elevation MI).

Outcomes: The primary outcome is difference in 30 day (plus/minus 5 days) occurrence of major adverse cardiac events (as defined later in this protocol) between placebo and Tocilizumab treated groups. Secondary outcomes to be assessed include length of hospitalization, readmission rates by day 30, CRP levels at 0 hours, 24 hours, 48 hours, and 30 days following treatment, and safety of Tocilizumab with focus on rates of known side effects.

DETAILED DESCRIPTION:
Interleukin 6 (IL-6) is a cytokine that has a pro-inflammatory effect on the immune system. Cytokines are a broad and loose category of small proteins (~5-20 kDa) that are important in cell signaling - they are released by cells and affect the behavior of other cells, and sometimes the releasing cell itself. IL-6 is an important mediator of fever and of the acute phase response. IL-6 is responsible for stimulating acute phase protein synthesis as well as the production of neutrophils in the bone marrow. The acute-phase response is the detectable change in acute phase proteins, a class of proteins whose plasma concentrations increase or decrease in response to inflammation. IL-6 is secreted by T cells and macrophages to stimulate the immune response during infection and after trauma, especially burns or other tissue damage leading to inflammation. Smooth muscle cells in the tunica media of many blood vessels also produce IL-6 as a pro-inflammatory cytokine. IL-6 is capable of crossing the blood-brain barrier and triggering production of Prostaglandin E2 in the hypothalamus, thereby changing the body's temperature set point. In muscle and fatty tissue, IL-6 stimulates energy mobilization that leads to increased body temperature. IL-6 can be secreted by macrophages in response to specific microbial molecules, referred to as pathogen-associated molecular patterns (PAMPs). IL-6 is also produced by adipocytes and is thought to be a reason why obese individuals have higher endogenous levels of CRP. IL-6 signals through a cell-surface type I cytokine receptor complex consisting of the ligand-binding IL-6Rα chain (CD126) and the signal-transducing component gp130 (also called CD130). CD130 is the common signal transducer for several cytokines but the expression of CD126 is restricted to certain tissues. As IL-6 interacts with its receptor, it triggers the gp130 and IL-6R proteins to form a complex, thus activating the receptor. These complexes bring together the intracellular regions of gp130 to initiate a signal transduction cascade through certain transcription factors.

Acute Myocardial Infarction (MI) occurs when myocardial ischemia, a diminished blood supply to the heart muscle, exceeds a critical threshold and overwhelms myocardial cellular repair mechanisms designed to maintain normal function. Ischemia at this critical threshold level for an extended period results in irreversible myocardial cell damage or death. A common clinical diagnostic classification scheme is based on electrocardiographic findings as a means of distinguishing between two types of acute MI, one that is marked by ST elevation (STEMI) and one that is not (NSTEMI). In acute MI IL-6 levels rapidly increase in response to ischemia and inflammation. In one study, plasma IL-6 levels were increased at all sampling points from admission to discharge in patients with acute MI as compared with IL-6 levels in controls. Cardiac catheterization did not influence plasma IL-6 levels. In another study, patients with acute MI demonstrated a peak in IL-6 levels on days 1 and 2 which then declined rapidly to lower, although not normalized, levels during hospitalization and at 6 and 12 weeks. It has also been demonstrated that elevated levels of IL-6 are associated with worse outcomes in acute MI. In one study elevated IL-6 levels at day 1 and day 30 were independent predictors of adverse events. In another study, on univariante analyses, baseline IL-6 was related to death but not recurrent non-fatal acute coronary syndromes. Another study demonstrated significant correlations between increased IL-6 levels and impaired left ventricle systolic and diastolic function supportive of a role of IL-6 in post-infarction cardiac damage. This same group also demonstrated that an increased level of IL-6 in acute MI was an independent predictor of left ventricle systolic and diastolic dysfunction 6 months after MI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 years old
* Subjects who present to Keesler Medical Center with clinical, physical examination, serologic, and electrocardiographic evidence of an acute MI (NSTEMI or STEMI), as determined by the treating physician

Exclusion Criteria:

* Subjects with clinical, physical examination, or radiographic evidence suspicious for active Tuberculosis (TB)
* Subjects with a known history of Hepatitis B or Hepatitis C infection This exclusion refers specific subjects who are actively being treated with medications for Hepatitis B or C or who have known virologic evidence on ongoing infection with Hepatitis B or C
* Subjects who are immune compromised including transplant recipients, patients with HIV, etc.
* Subjects with evidence of Tuberculosis infection on chest xray
* Subjects with known allergic reaction to tocilizumab or other IL-6 inhibitors
* Subjects with clinical, physical examination, serologic, or radiographic evidence of active infection
* Subjects receiving therapy for malignancy-this will not exclude subjects receiving therapy for non-melanoma skin cancer such as basal cell carcinoma or squamous cell carcinoma of the skin
* Female subjects who are pregnant or breast-feeding
* Subjects with existing cognitive impairment such as known moderate to severe dementia or subjects who present with new onset delirium

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Carroll, MD, Principal Investigator — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States

REFERENCES:
- [Derived] Carroll MB, Haller C, Smith C. Short-term application of tocilizumab during myocardial infarction (STAT-MI). Rheumatol Int. 2018 Jan;38(1):59-66. doi: 10.1007/s00296-017-3842-y. Epub 2017 Oct 24. PMID 29067495

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab | Placebo
Started | 12 | 16
Completed | 11 | 16
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data as well as medication use, type of MI recorded
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Categorical [Count of Participants; unit: Participants] — Age at the time of enrollment
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 9 | 12
    >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (10.0) | 67.7 (9.5) | 69.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 14 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American (Black) | 0 | 1 | 1
  Caucasian (White) | 12 | 13 | 25
  Hispanic | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants] — Demographics of study participants
  Participants
    United States | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Cardiovascular Events (MACE)
Description: 30 day rate of major adverse cardiac events (MACE) following administration of Tocilizumab subcutaneously single dose within 24 hours of NSTEMI or STEMI as compared to administration of placebo
Time Frame: 30 days after one time injection
Population: Major Adverse Cardiac Events (MACE) for those gathered 30 days after receiving medication or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 9 | 3
Participants
  Death | 0 | 0
  Recurrent Myocardial Infarction | 2 | 1
  Dysrhythmia | 2 | 1
  Septal/Valve Rupture | 1 | 1
  Pericarditis | 2 | 0
  Cardiac Tamponade | 2 | 0

ADVERSE EVENTS:
Time Frame: Major adverse cardiac event (MACE) rate consisting of several outcomes reported herein were collected 30 days after enrollment
Description: Information was collected from direct assessment, follow-up phone interview, and record review.
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/16
Other Adverse Events (participants affected / at risk) | 0/11 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=11) | Placebo (N=16)
Symptomatic bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Heart rate below 60 beats per minute, not due to beta-blocker or calcium channel blocker use.
Symptomatic Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Systolic blood pressure below 90 mm Hg not due to medication with symptoms
Gross Hematuria (General disorders) | 1 (1) | 0 (0) — Frank blood in the urine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-09-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT02419937/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02419937/ICF_001.pdf